CLINICAL TRIAL: NCT00923962
Title: Endothelial and Metabolic Effects of GLP-1 in Coronary Circulation in Patients With Type 2 Diabetes Mellitus
Brief Title: Endothelial and Metabolic Effects of Glucagon-like Peptide-1 (GLP-1) in Coronary Circulation in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jacob Christian Sivertsen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLP-1 Coronary circulation 01
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Basic science; Type 2 Diabetes mellitus; Glucagon like peptid-1; Coronary Bloodflow; Metabolite uptake
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 2 Diabetes patients (Active Comparator)
  Interventions: Drug: Glucagon like peptide-1; Drug: Adenosine
- Healthy (Active Comparator)
  Interventions: Drug: Glucagon like peptide-1; Drug: Adenosine
- Artherosclerosis (Active Comparator)
  Interventions: Drug: Glucagon like peptide-1; Drug: Adenosine

INTERVENTIONS:
Drug: Glucagon like peptide-1 — 0,1 pmol/kg/min
Drug: Adenosine — 20-40 microgram/minute

SUMMARY:
GLP-1 is an incretin hormone which is discharged from the intestines after food intake. The hormone is known for its powerful insulinotropic and trophic effects on the beta cells in the pancreas and is currently used as an anti-diabetic agent in patients with type 2 diabetes (T2DM).

GLP-1 receptors are widely distributed including on the endothelial cells in both coronary and skeletal muscle circulation and on the myocardium. GLP-1-receptor studies on knock-out mice have shown that they exhibit a reduced myocardial contractility and reduced diastolic heart function. GLP-1 also shows beneficial cardiovascular effects in patients with acute myocardial infarctions and dogs with dilated cardiomyopathy in that the left ventricle function and endothelial dysfunction improves after GLP-1 treatment via insulin-independent mechanisms. Preclinical studies indicate that exogenous administrated GLP-1 in physiological concentrations can improve perfusion but this has never been tested in humans. It is also unknown whether GLP-1 can directly increase the glucose/metabolite uptake across both cardiac and skeletal muscle in an insulin independent manner. Unpublished studies do however indicate that the improvement in the cardiovascular system is largely dependent upon a high blood glucose level and only partially dependent upon the antiglycemic effects of GLP-1.

In the proposed studies the investigators wish to examine the physiological role of GLP-1 receptor stimulation both with regard to perfusion, metabolic improvement as well as cardiac inotropic. These studies will be conducted in both healthy and in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians over 18
* Emitted for non-acute coronary arteriography (CAG) in Gentofte hospital
* BMI 23-35 kg/m2
* Normal hemoglobin
* Who gives informed consent
* Those with type 2 diabetes: HbA1c 6-10%
* Those without type 2 diabetes: Normal oral glucose tolerance test (OGTT) according to WHO criteria

Exclusion Criteria:

* Liver disease (ALAT > 2x normal)
* Diabetic nefropati (Creatinine > 130 µM or albuminuria)
* Treatment with medicine that cannot be paused 12 hours before intervention
* Pregnancy or breastfeeding
* Insulin- or glitazone treatment
* Healthy controls: close family history with diabetes
* Unstable angina pectoris
* Non-STEMI
* Atrial fibrillation
* Valvular disease
* LVEF < 50%
* Severe systemic disease
* Type 1 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Coronary blood flow | 10 minutes after I.A. GLP-1
Coronary metabolite uptake | 10 minutes after I.A. GLP-1

CONTACTS AND LOCATIONS:
Overall Officials: Jan S Jensen, MD, DMSc, Study Chair — University hospital Gentofte, Department of Cardiology; Jaya Rosenmeier, MD, Ph.D., Principal Investigator — University hospital Gentofte, Department of Cardiology
Locations (1):
- University Hospital Gentofte, Department of Cardiology, Gentofte Municipality, Denmark

REFERENCES:
- [Background] Bjallmark A, Larsson M, Winter R, Westholm C, Jacobsen P, Lind B, Brodin LA. Velocity tracking--a novel method for quantitative analysis of longitudinal myocardial function. J Am Soc Echocardiogr. 2007 Jul;20(7):847-56. doi: 10.1016/j.echo.2006.11.024. PMID 17617311
- [Background] Diamant M, Lamb HJ, Groeneveld Y, Endert EL, Smit JW, Bax JJ, Romijn JA, de Roos A, Radder JK. Diastolic dysfunction is associated with altered myocardial metabolism in asymptomatic normotensive patients with well-controlled type 2 diabetes mellitus. J Am Coll Cardiol. 2003 Jul 16;42(2):328-35. doi: 10.1016/s0735-1097(03)00625-9. PMID 12875772
- [Background] Edwards CM, Todd JF, Mahmoudi M, Wang Z, Wang RM, Ghatei MA, Bloom SR. Glucagon-like peptide 1 has a physiological role in the control of postprandial glucose in humans: studies with the antagonist exendin 9-39. Diabetes. 1999 Jan;48(1):86-93. doi: 10.2337/diabetes.48.1.86. PMID 9892226
- [Background] Golpon HA, Puechner A, Welte T, Wichert PV, Feddersen CO. Vasorelaxant effect of glucagon-like peptide-(7-36)amide and amylin on the pulmonary circulation of the rat. Regul Pept. 2001 Dec 15;102(2-3):81-6. doi: 10.1016/s0167-0115(01)00300-7. PMID 11730979
- [Background] Luque MA, Gonzalez N, Marquez L, Acitores A, Redondo A, Morales M, Valverde I, Villanueva-Penacarrillo ML. Glucagon-like peptide-1 (GLP-1) and glucose metabolism in human myocytes. J Endocrinol. 2002 Jun;173(3):465-73. doi: 10.1677/joe.0.1730465. PMID 12065236
- [Background] Mogelvang R, Sogaard P, Pedersen SA, Olsen NT, Schnohr P, Jensen JS. Tissue Doppler echocardiography in persons with hypertension, diabetes, or ischaemic heart disease: the Copenhagen City Heart Study. Eur Heart J. 2009 Mar;30(6):731-9. doi: 10.1093/eurheartj/ehn596. Epub 2009 Jan 27. PMID 19176536
- [Background] Nichols GA, Hillier TA, Erbey JR, Brown JB. Congestive heart failure in type 2 diabetes: prevalence, incidence, and risk factors. Diabetes Care. 2001 Sep;24(9):1614-9. doi: 10.2337/diacare.24.9.1614. PMID 11522708
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Background] Yu M, Moreno C, Hoagland KM, Dahly A, Ditter K, Mistry M, Roman RJ. Antihypertensive effect of glucagon-like peptide 1 in Dahl salt-sensitive rats. J Hypertens. 2003 Jun;21(6):1125-35. doi: 10.1097/00004872-200306000-00012. PMID 12777949
- [Background] Nystrom T, Gutniak MK, Zhang Q, Zhang F, Holst JJ, Ahren B, Sjoholm A. Effects of glucagon-like peptide-1 on endothelial function in type 2 diabetes patients with stable coronary artery disease. Am J Physiol Endocrinol Metab. 2004 Dec;287(6):E1209-15. doi: 10.1152/ajpendo.00237.2004. Epub 2004 Sep 7. PMID 15353407
- [Background] Bullock BP, Heller RS, Habener JF. Tissue distribution of messenger ribonucleic acid encoding the rat glucagon-like peptide-1 receptor. Endocrinology. 1996 Jul;137(7):2968-78. doi: 10.1210/endo.137.7.8770921.
- [Background] Wei Y, Mojsov S. Tissue-specific expression of the human receptor for glucagon-like peptide-I: brain, heart and pancreatic forms have the same deduced amino acid sequences. FEBS Lett. 1995 Jan 30;358(3):219-24. doi: 10.1016/0014-5793(94)01430-9. PMID 7843404
- [Background] Wei Y, Mojsov S. Distribution of GLP-1 and PACAP receptors in human tissues. Acta Physiol Scand. 1996 Jul;157(3):355-7. doi: 10.1046/j.1365-201X.1996.42256000.x. No abstract available. PMID 8830893
- [Background] Nikolaidis LA, Elahi D, Shen YT, Shannon RP. Active metabolite of GLP-1 mediates myocardial glucose uptake and improves left ventricular performance in conscious dogs with dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2005 Dec;289(6):H2401-8. doi: 10.1152/ajpheart.00347.2005. Epub 2005 Jul 15. PMID 16024574
- [Background] Ban K, Noyan-Ashraf MH, Hoefer J, Bolz SS, Drucker DJ, Husain M. Cardioprotective and vasodilatory actions of glucagon-like peptide 1 receptor are mediated through both glucagon-like peptide 1 receptor-dependent and -independent pathways. Circulation. 2008 May 6;117(18):2340-50. doi: 10.1161/CIRCULATIONAHA.107.739938. Epub 2008 Apr 21. PMID 18427132
- [Background] Nystrom T, Gonon AT, Sjoholm A, Pernow J. Glucagon-like peptide-1 relaxes rat conduit arteries via an endothelium-independent mechanism. Regul Pept. 2005 Feb 15;125(1-3):173-7. doi: 10.1016/j.regpep.2004.08.024. PMID 15582729